CLINICAL TRIAL: NCT02907905
Title: Epidemiology of Hepatitis A,B and C Virus by Dried Blood Spot in Homeless Population
Brief Title: Epidemiology of Viral Hepatitis Among Subjects in Precarious
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9609
Record Dates: First submitted 2016-09-12; First posted 2016-09-20 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Social Insecurity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Population homeless or living in slum (Other): Population homeless or living in slum realizing realizing a capillary sampling
  Interventions: Biological: capillary sampling

INTERVENTIONS:
Biological: capillary sampling — After elution in buffer (PBS-Tween azide and thiamol) eluate 200 microliter is processed on automated techniques (Siemens Centaur XL and Diasorin) after adjustment of the figures according to ISO 15189 scope B.
  The results are qualitatively made and sent to the teams. The return of results, a proposal for appropriate care in the event of contact with virus (anti-HAV HCV HBV) through a rendering consultation results

SUMMARY:
Social insecurity is a significant cost in human terms (health and societal), it defines evil and can be identified as difficulties accessing health and especially water.

We chose to take stock of these populations defined by difficulties accessing water as precarious setting. Subjects homeless population fall into this by accident of life, a life "homeless" or migrant subjects often illegally having only transitory access (associative or charitable structures host) the conditions precarious sanitation including drinking water or toilet. Populations of slums in the same conditions or the presence rationed water (one tap for 150 people) restricts hygiene.

DETAILED DESCRIPTION:
Social insecurity is a significant cost in human terms (health and societal), it defines evil and can be identified as difficulties accessing health and especially water.

We chose to take stock of these populations defined by difficulties accessing water as precarious setting. Subjects homeless population fall into this by accident of life, a life "homeless" or migrant subjects often illegally having only transitory access (associative or charitable structures host) the conditions precarious sanitation including drinking water or toilet. Populations of slums in the same conditions or the presence rationed water (one tap for 150 people) restricts hygiene.

The sampling system as part of a consultation in routine care (will be in DBS (blotter) only alternative to invasive venous sample and requiring heavier care facility. The capillary sampling on filter will also detect a marker of malnutrition .

Thus in live in large social precariousness adult this study should show which interventions in public health and management proposals are most appropriate for this population.

ELIGIBILITY:
Inclusion Criteria:

* Population homeless (SDF)
* Population living in slums.

Exclusion Criteria:

* Pregnant or lactating women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
serology HBV | 1 day
  Study prevalence HBV in these precarious populations
serology HCV | 1 day
  Study prevalence HCV in these precarious populations
serology HAV | 1 day
  Study prevalence HAV in these precarious populations

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Ducos, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- DUCOS, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided